CLINICAL TRIAL: NCT02399293
Title: Computer-based Attention Training in Patients With Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Hammel Neurocenter (Other)
Responsible Party: Principal Investigator, Jonas Lindeløv, M.sc., Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hnrc_nback
Record Dates: First submitted 2015-03-11; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Brain Injuries
Keywords: Cognitive training; Cognitive rehabilitation; Acquired brain injury; N-back; Visual Search; Cognitive transfer
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Patient N-back (Experimental): Patients training the N-back task
  Interventions: Behavioral: N-back
- Patient Visual Search (Active Comparator): Patients training the Visual-Search task
  Interventions: Behavioral: Visual Search
- Non-impaired N-back (Experimental): Non-impaired training the N-back task
  Interventions: Behavioral: N-back
- Non-impaired Visual Search (Active Comparator): Non-impaired training the Visual-Search task
  Interventions: Behavioral: Visual Search

INTERVENTIONS:
Behavioral: N-back — The N-back task required patients to monitor a continuous sequence of stimuli (in this experiment audio and visual stimuli). Press a button if the current stimulus is the same as that shown N back in the sequence. N increases if performance is good and decreases if performance is poor.
  Subjects train for 20 days, 12 blocks a day, 20+N trials per block. That is 240 blocks in total. A minimum of 10 blocks per day counts as a successfully trained day.
  Arms: Non-impaired N-back; Patient N-back
Behavioral: Visual Search — The Visual Search task consists of a NxN array of shapes. Press the button if a certain target stimulus is present in this array. N increases if performance is good and decreases if performance is poor.
  Subjects train for 20 days, 12 blocks a day, 20+N trials per block. That is 240 blocks in total. A minimum of 10 blocks per day counts as a successfully trained day.
  Arms: Non-impaired Visual Search; Patient Visual Search

SUMMARY:
Investigates computer based cognitive rehabilitation and training using the N-back task with a Visual Search task as an active control. The overall purpose is to provide (further) evidence about the efficacy (or lack of efficacy) of the N-back task and to find points of convergence and divergence between patients with acquired brain injury and non-impaired subjects.

ELIGIBILITY:
Inclusion criteria:

* subjects should be able to do both task at level at the time of recruitment
* Informed consent
* (for brain injured patients) training must not interfere with treatment as usual.
* (for brain injured patients) no symptoms which hinder testing and training. I.e. aphasia, deafness, tetraplegia etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline Raven's advanced progressive matrices at the end of training | within five days after 20 full training days has been completed. Expected 3-6 weeks after baseline.

SECONDARY OUTCOMES:
Change from baseline WAIS-III Working Memory Index at the end of training | within five days after 20 full training days has been completed. Expected 3-6 weeks after baseline.
Change from baseline WAIS-III Processing Speed Index at the end of training | within five days after 20 full training days has been completed. Expected 3-6 weeks after baseline.
Change from baseline Operation Span at the end of training | within five days after 20 full training days has been completed. Expected 3-6 weeks after baseline.
Change from baseline Stroop color-text interference at the end of training | within five days after 20 full training days has been completed. Expected 3-6 weeks after baseline.
Change from baseline AMPS at the end of training | within five days after 20 full training days has been completed. Expected 3-6 weeks after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Lindeløv, M.Sc., Principal Investigator — Hammel Neurocenter